CLINICAL TRIAL: NCT03918382
Title: Management of Side Effects in Head and Neck Cancer by Systematic Use of PRO During Radiotherapy- The National DAHANCA PRO Study
Brief Title: Patient-Reported Outcomes in Head and Neck Cancer
Acronym: DAHANCA PRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Comprehensive Cancer Center (Other); Danish Cancer Society (Other); University of Copenhagen (Other); Danish Head and Neck Cancer Group (Network); Herlev Hospital (Other); Zealand University Hospital (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Helle Pappot, Clinical Oncologist, Consultant, DMSc, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: DAHANCA PRO
Record Dates: First submitted 2019-04-10; First posted 2019-04-17 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Cancer; Radiotherapy Side Effect
Keywords: Patient-Reported Outcome; Quality of life; Electronic reporting of symptoms; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: A prospective nation-wide, sequential cohort study.
  * First phase control group. 97 participants. No Intervention: Standard of care.This arm will continue standard procedure regarding side effect registration and handling.
  * Second phase. PRO group. 194 participants. Intervention: Active use of electronic patient-reported outcomes.This arm will be assigned to intervention by weekly electronic reporting of side effects and quality of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): First phase. 97 participants. This group will continue standard procedure regarding side effect registration and handling. When the 97 patients have been included and have finished their radiotherapy the second phase will be initiated.
- PRO group (Experimental): Second phase. 194 participants. This group will be assigned to the intervention which is weekly electronic Patient-Reported Outcomes. Patients report the symptoms (PRO) on a tablet before each weekly control visit. The clinician will use the patients PRO answers as part of the consultation. The PRO symptoms consist of head and neck relevant items fra PRO-CTCAE™ (Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) and EORTC (European Organisation for Research and Treatment of Cancer) item library.
  Interventions: Other: Electronic Patient-Reported Outcome

INTERVENTIONS:
Other: Electronic Patient-Reported Outcome — Weekly reporting of patient-reported outcomes on a tablet for closer contact between patient and clinic during radiotherapy.
  Other Names: Real-time guidance of patients when symptom reporting; Patient Self-Reporting of Symptoms
  Arms: PRO group

SUMMARY:
Weekly electronic reporting of patient-reported outcomes will be tested in a national trial in participants undergoing radiotherapy for head and neck cancer.

The study is a national study under the Danish Head and Neck Cancer Group (DAHANCA) and all 6 centers in Denmark will participate.

The clinical endpoints will be:

* Quality of life
* Objective toxicity score (DAHANCA)
* Opioid treatment
* Tube feeding
* Weight loss
* Hospitalization
* Compliance to treatment

DETAILED DESCRIPTION:
There is a high level of evidence for improved disease control in head and neck cancer (HNC) using regimens with accelerated radiotherapy and concomitant chemotherapy. These intense regimens can result in severe acute and late side effect. The standard approach for documenting symptomatic adverse events (AEs) in cancer clinical trials involves investigator reporting using the National Cancer Institute's (NCI's) Common Terminology Criteria for Adverse Events (CTCAE). In Denmark, the Danish Head and Neck Cancer Group (DAHANCA) toxicity score has been used as an instrument in assessing objective treatment induced toxicity. New research in other cancer treatments indicate, that systematic patient assessment of side effects may improve treatment outcome. Patient Reported Outcomes (PROs) can be used for symptom monitoring. Interactive use of PRO may secure early recognition of specific symptoms in the individual patient and timely management of side effects.

This trial it is a prospective nationwide, single armed sequential cohort study will investigate the effects of active use of PROs in clinical counselling and decision making during primary or post-operative curative radiotherapy for squamous-cell carcinoma of the head and neck (HNSCC). It will investigate quality of life and the management of side effects in standard clinical counselling (control group) versus standard clinical counselling plus the PRO (PRO group). The EORTC QLQ-C30 (quality of life questionnaire) and EQ-D5-L5 will be answered in both groups. In the PRO group the participants will be asked to complete the electronic PRO (PRO CTCAE™ HNC relevant items supplemented by HNC specific items fra the EORTC library) weekly. The electronic PRO questionnaire is designed to give feedback to treating physician and nurses at visits during and shortly after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary or post-operative curative radiotherapy (photons) plus/minus concomitant Cisplatinum for squamous-cell carcinoma of the head and neck (HNSCC)
* No serious cognitive deficits
* Read and understand Danish

Exclusion Criteria:

•Prior radiotherapy in the same area (head and neck)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life measured by EORTC QLQ C30 | With in the first 2 months
  Registration of differences in quality of life between the two groups in the study. EORTC QLQ-C30(scale range 0-100, a higher score indicating better quality of life) will be used for as quality of life measurement. The scores will be presented graphically in separate figures. Differences between the groups will be tested using t-test and analysis of covariance.
Quality of life (QOL) measured by EuroQol EQ-5D-5L. | With in the first 2 months
  EQ-5D-5L measures individual generic health status using 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each dimension has 5 levels depending on severity of symptoms (1 no problems, 5 extreme problems) and a VAS (visual analogue scale). The scores can then be converted into a single index number. The index value will be used for calculation of quality-adjusted life years (QALYs) for a health economic analysis of the intervention. The scores will be presented graphically in separate figures. Differences between the groups will be tested using t-test and analysis of covariance.

SECONDARY OUTCOMES:
DAHANCA toxicity score | Within the first 4 months
  DAHANCA toxicity score is an objective grading of the patients symptoms by the clinician. Scale 0-4, where 0 is no/nothing and 4 is severe. Registration of differences in DAHANCA toxicity score and electronic PRO
Weight loss | Within the first 4 months
  Registration of differences in weight loss in the two groups.
Hospitalization due to toxicity expect tube-feeding and patients reported experience | Within the first 4 months
  Number of hospitalizations reported in the medical record at the control visit 2 months after end af radiotherapy
Compliance to cisplatinum | Within the first 2 months
  Number of participants completing planned Cisplatinum
Time to opioid treatment | Within the first 3 months
  Registration of differences in time to opioid treatment in the two groups
Time to tube-feeding/other feeding | Within the first 3 months
  Registration of differences in time to Time to tube-feeding/other feeding in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Holländer-Mieirtz, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Copenhagen
  - Rigshoapitalet, Copenhagen
  - Zealand Hospital, Næstved
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study protocol article — https://pubmed.ncbi.nlm.nih.gov/32056473/